CLINICAL TRIAL: NCT05988723
Title: Evaluation of the Effects of Obesity on Orthodontic Tooth Movement
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Mustafa UZUN, Research Assistant, Aydin Adnan Menderes University
Other Study IDs: DHF-21006
Record Dates: First submitted 2023-06-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Obesity, Childhood; Orthodontic Treatment
Keywords: Obesity; Orthodontic Treatment; Tooth movement; Biomarkers
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group (obese patient): Leptin, IL-6, OPG, RANKL levels were measured in samples taken from the distal gingival groove of the canine teeth of obese individuals. Roth metal brackets and tubes with 0.022 inch slots were used for the fixed orthodontic treatment of the patients. After leveling the teeth of the patients with arch wires, it was waited for 2 months in 19x25 stainless steel arch wire and then 150 gr distalization force was applied. DOS samples were taken from the distal gingival groove of teeth on day 7 (T2), day 14 (T3) and day 21 (T4), just before distalization force was applied (T0), 24 hours after force was applied (T1). In order to determine the speed of tooth movement, the patient's mouth was scanned on the days when DOS was taken (T0,T1,T2,T3,T4) and in addition to these days, on the 28th day (T5) and at the end of the 3rd month (T6), and the amount of movement of the canine tooth was measured in mm. Leptin, IL-6, OPG, RANKL levels were examined with Elisa kits from the samples obtained.
  Interventions: Other: ELISA kits
- Control Group (normal patient): Leptin, IL-6, OPG, RANKL levels were measured in samples taken from the distal gingival groove of the canine teeth of normal weight individuals.Roth metal brackets and tubes with 0.022 inch slots were used for the fixed orthodontic treatment of the patients.After leveling the teeth of the patients with arch wires, it was waited for 2 months in 19x25 stainless steel arch wire and then 150 gr distalization force was applied.DOS samples were taken from the distal gingival groove of teeth on day 7 (T2), day 14 (T3) and day 21 (T4), just before distalization force was applied (T0), 24 hours after force was applied (T1). In order to determine the speed of tooth movement, the patient's mouth was scanned on the days when DOS was taken (T0,T1,T2,T3,T4) and in addition to these days, on the 28th day (T5) and at the end of the 3rd month (T6), and the amount of movement of the canine tooth was measured in mm. Leptin, IL-6, OPG, RANKL levels were examined with Elisa kits from the samples obtained.
  Interventions: Other: ELISA kits

INTERVENTIONS:
Other: ELISA kits — Making biochemical measurements with the ELISA kit

SUMMARY:
In this study, bone remodeling in the gingival crevicular fluid was evaluated biochemically during canine distalization in obese individuals and compared with normal weight individuals. At the same time, the speed of tooth movement was measured in obese individuals and compared with normal weight individuals.

DETAILED DESCRIPTION:
Among the obese and normal weight patients who applied to Aydın Adnan Menderes University Faculty of Dentistry Department of Orthodontics for orthodontic treatment, those who met the inclusion criteria were selected for the study. Patients with Angle Class II malocclusion who required extraction of the maxillary first premolar tooth were included in the study. Obesity classification, as the World Health Organization (WHO) determines the obesity values in children; BMI values; <5% very thin, 5%-15% underweight, 16-85% normal, 86-95% overweight, and ≥95% obese. Percentile values were calculated with reference to the study "Reference Values for Weight, Height, Head Circumference, and Body Mass Index in Turkish Children" conducted by Neyzi et al. (2015). In our study, individuals with normal weight and without any systemic disease were determined as the control group, and individuals without any systemic disease other than obesity were determined as the study group. Leptin, IL-6, OPG and RANKL levels were measured in gingival sulcus fluid samples taken from the distal gingival groove of obese and healthy individuals who underwent canine distalization. Roth metal brackets and tubes with 0.022 inch slots were used for the fixed orthodontic treatment of the patients. After leveling the teeth of the patients with arch wires, it was waited for 2 months in 19x25 stainless steel arch wire and then 150 gr distalization force was applied. DOS samples were taken from the distal gingival groove of teeth on day 7 (T2), day 14 (T3) and day 21 (T4), just before distalization force was applied (T0), 24 hours after force was applied (T1). In order to determine the speed of tooth movement, the patient's mouth was scanned on the days of DOS (T0, T1, T2, T3, T4) and in addition to these days, on the 28th day (T5) and at the end of the 3rd month (T6), with the 3shape Trios device and using the OrthoAnalyzer software. The amount of movement of the canine tooth was measured in mm. Before collecting the gingival groove fluid sample, the area was isolated with cotton rolls, and the adjacent teeth and marginal gingival area were air-dried. The Periopaper was then gently placed in the gingival sulci below the gingival margin for 30 seconds. Paper strips were individually sealed in eppendorf tubes and each sample was stored at -80°C until later analysis. Leptin, IL-6, OPG and RANKL levels were examined with Elisa kits from the samples obtained. The planned period for the study was determined as 3 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 95% for obese individuals, body mass index between 16-85% for normal weight individuals,
* Absence of any systemic disease that may affect tooth movement,
* Premolar tooth extraction is required because the patients have Angle Class II malocclusion,
* No history of orthodontic treatment,
* No anti-inflammatory drug use within 1 month before starting the study,
* No signs of gingivitis or a history of periodontal treatment,
* To have good periodontal health,
* The patients are in the permanent dentition period,

Exclusion Criteria:

* History of previous orthodontic treatment,
* Anti-inflammatory drug use within 1 month before starting the study,
* To have signs of gingivitis or a history of periodontal treatment,
* Individuals with poor periodontal health,
* Individuals in the mixed dentition period,
* Individuals who have smoking or alcohol habits,
* Determined as patient non-compliance.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Men and women patients aged between 12-18 years who have continued orthodontic treatmens
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Leptin, RANKL, OPG and IL-6 ELISA kits | The change in biomarker levels will be measured over a 1-month period.
  ELISA kits were used to measure the biomarker level in gingival crevicular fluid samples taken from the patient.
Correlation between leptin level and tooth movement speed | It will be examined whether there is a relationship between leptin level and tooth movement speed over a 21-day period.
  3D intraoral scanner and leptin elisa kit will be used

CONTACTS AND LOCATIONS:
Overall Officials: Mine Geçgelen Cesur, Study Director — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University Faculty of Dentistry, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dilsiz A, Kilic N, Aydin T, Ates FN, Zihni M, Bulut C. Leptin levels in gingival crevicular fluid during orthodontic tooth movement. Angle Orthod. 2010 May;80(3):504-8. doi: 10.2319/072109-402.1. PMID 20050744
- [Result] Neyzi O, Bundak R, Gokcay G, Gunoz H, Furman A, Darendeliler F, Bas F. Reference Values for Weight, Height, Head Circumference, and Body Mass Index in Turkish Children. J Clin Res Pediatr Endocrinol. 2015 Dec;7(4):280-93. doi: 10.4274/jcrpe.2183. PMID 26777039
- [Result] Jayachandran T, Srinivasan B, Padmanabhan S. Salivary leptin levels in normal weight and overweight individuals and their correlation with orthodontic tooth movement. Angle Orthod. 2017 Sep;87(5):739-744. doi: 10.2319/120216-869.1. Epub 2017 May 4. PMID 28471265
- [Result] Saloom HF, Boustan R, Seehra J, Papageorgiou SN, Carpenter GH, Cobourne MT. The impact of obesity on orthodontic treatment outcome in adolescents: a prospective clinical cohort study. Eur J Orthod. 2021 Apr 3;43(2):165-172. doi: 10.1093/ejo/cjaa032. PMID 32390057